CLINICAL TRIAL: NCT04223388
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Research Study to Investigate the Safety and Efficacy of a Probiotic Lactobacillus Plantarum 276 (Lp276) on Gastrointestinal Health in Healthy Adults
Brief Title: A Study to Investigate the Safety and Efficacy of a Probiotic on Gastrointestinal Health in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Church & Dwight Company, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19PGHC
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Health; Healthy
Keywords: Probiotics; Healthy; Gut Health; Gastrointestinal Health

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Lactobacillus plantarum 276
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum 276 — 5 Billion CFU/dose, serving size = 1 capsule/day
  Other Names: Lp276
  Arms: Probiotic
Other: Placebo — Placebo product, serving size = 1 capsule/day
  Arms: Placebo

SUMMARY:
Eligible participants will be randomized and receive either the probioic or placebo supplement to consume daily for 28-days. Three check-in visits will occur every 7 days of study participation. Participants will be expected to complete a daily study diary documenting their investigational product use/adverse events and a daily bowel habits diary documenting each bowel movement. Blood samples, stool samples, and questionnaires will be completed for study outcome analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males between 18 to 55 years of age, inclusive
2. BMI between 18.5 to 32 kg/m2, inclusive
3. Self-reported history of diarrhea over the last 3 months, defined as > 5 BMs with the majority (≥ 50%) of the BMs per week being Bristol stool form types ≥5, 6 or 7
4. Female participant is not of child bearing potential, which is defined as females who have had a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation, or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR,

   Females of childbearing potential must agree to use a medically approved method of birth control and must have negative urine pregnancy test results at screening and baseline. A minimum of 3-months stable dose is required for females on a hormonal birth control. Acceptable methods of birth control include:

   I. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System) II. Double-barrier method III. Intrauterine devices IV. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s) V. Vasectomy of partner (shown successful as per appropriate follow-up)
5. Healthy as determined by laboratory results, medical history and physical exam by QI
6. Agrees to comply with all study procedures
7. Agrees to refrain from the use of any home remedies to control GI issues if live bacteria may be involved
8. Agrees to avoid NSAIDs and Steroids for 72 hours and Vitamin C and related supplements for 24 hours prior to fecal zonulin sample collection
9. Agrees to maintain current level of physical activity and diet throughout the study
10. Agrees to provide written informed consent

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Allergy or sensitivity to investigational product's active or inactive ingredients
3. Clinically significant abnormal laboratory results at screening as assessed by QI
4. Chronic use of anti-diarrhea medications and supplements; occasional use is permitted based on frequency of use and appropriate wash-out to be determined by QI
5. Currently undergoing pharmacological treatment for IBS, or history of active treatment for IBS within the last 1 year
6. Clinically significant disease of the gastrointestinal tract (examples include but are not limited to celiac disease, gluten intolerance/sensitivity, inflammatory bowel disease)
7. Gastrointestinal surgery within the past 3 months. Gastrointestinal surgery > 3 months ago, will be assessed by the QI on a case-by-case basis.
8. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Minor surgery will be considered on a case by case basis by QI
9. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Cancer in full remission for more than five years after diagnosis are acceptable.
10. Verbal confirmation of autoimmune disease or if immune-compromised
11. Verbal confirmation of HIV, hepatitis B/C positive diagnosis
12. Metabolic syndrome or chronic diseases to be assessed by QI on a case by case basis
13. Type I or Type II diabetes
14. Significant cardiovascular event in the past 6 months. No significant cardiovascular event on stable medication may be included after assessment by the QI on a case by case basis
15. History or currently with kidney and liver diseases assessed by QI on a case by case basis, with the exception of the history of kidney stones symptom-free for 1 year
16. Verbal confirmation of current or pre-existing thyroid condition. Treatment on a stable dose medication for over 6 months will be reviewed on a case-by-case basis by the QI
17. Blood or bleeding disorders, with the exception of a history of anemia caused by deficiency of a mineral or vitamin, and no longer present
18. Current use or consumption of antibiotics in the 4 weeks prior to baseline
19. Current use or consumption of prebiotic or probiotic or synbiotic supplements in the 4 weeks prior to baseline
20. Current use of prescribed medications that may affect the study outcomes
21. Use of over-the-counter (OTC) medications or supplements or consumption of foods/drinks that may affect the study outcomes, unless willing to undergo an appropriate washout period prior to baseline is agreed upon after assessment by the QI
22. Use of medical marijuana
23. Chronic use of recreational marijuana; infrequent use (>30 days since last use) to be assessed by QI
24. Use of tobacco products unless quit 90 days prior to baseline
25. Alcohol or drug abuse in the past year
26. High alcohol intake (average of >2 standard drinks per day or >10 standard drinks per week)
27. Use of narcotics
28. Illicit drug use in the past 6 months as assessed by the QI
29. Participation in other clinical research trials 30 days prior to randomization or will be participating in another investigation during the study
30. Participants who plan to donate blood during the study or within 30 days of completing the study
31. Any known (choric or acute) medical or neuropsychological condition that, in the QI's opinion, could interfere with study participation, or individuals who are cognitively impaired and/or who are unable to give informed consent
32. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The difference between probiotic and placebo groups in the change in gastrointestinal health from baseline to day 28 as determined by stool frequency as per daily bowel habit diary | 28 days
  Number of bowel movements per day will be assessed in the bowel habits diary
The difference between probiotic and placebo groups in the change in gastrointestinal health from baseline to day 28 as determined by stool consistency as per the Bristol Stool Scale | 28 days
  Bristol Stool Scale is a seven-stool description and image scale within the Daily Bowel Habit Diary to assess stool shape and consistency (1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = like a sausage but with cracks on its surface, 4 = like a sausage or snake, smooth and soft, 5 = soft blobs with clear-cut edges, 6 = fluffy pieces with ragged edges/mushy stool, 7 = watery, no solid pieces).
The difference between probiotic and placebo groups in the change in gastrointestinal health from baseline to day 28 as determined by gastrointestinal (GI) symptoms as per the gastrointestinal symptom rating scale | 28 days
  The GSRS is a validated, self-assessed, disease-specific scale that will be administered at all in-clinic visits. Five symptom clusters depicted as Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation will be assessed from the combination of the 15 items in the questionnaire (Abdominal pains, Heartburn, Acid regurgitation, Sucking sensations in the epigastrium, Nausea and vomiting, Borborygmus, Abdominal distension, Eructation, Increased flatus, Decreased passage of stools, Increased passage of stools, Loose stools, Hard Stools, Urgent need for defecation, Feeling of incomplete evacuation). All the domains will be scored on a 3-point scale where 1 represented no symptoms and 3 represented severe symptoms

SECONDARY OUTCOMES:
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 7 as determined by stool frequency as per the daily bowel habits diary | 7 days
  Number of bowel movements per day will be assessed in the bowel habits diary
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 14 as determined by stool frequency as per the daily bowel habits diary | 14 days
  Number of bowel movements per day will be assessed in the bowel habits diary
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 21 as determined by stool frequency as per the daily bowel habits diary | 21 days
  Number of bowel movements per day will be assessed in the bowel habits diary
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 7 as determined by stool consistency as per the Bristol Stool Scale | 7 days
  Bristol Stool Scale is a seven-stool description and image scale within the Daily Bowel Habit Diary to assess stool shape and consistency (1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = like a sausage but with cracks on its surface, 4 = like a sausage or snake, smooth and soft, 5 = soft blobs with clear-cut edges, 6 = fluffy pieces with ragged edges/mushy stool, 7 = watery, no solid pieces).
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 14 as determined by stool consistency as per the Bristol Stool Scale | 14 days
  Bristol Stool Scale is a seven-stool description and image scale within the Daily Bowel Habit Diary to assess stool shape and consistency (1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = like a sausage but with cracks on its surface, 4 = like a sausage or snake, smooth and soft, 5 = soft blobs with clear-cut edges, 6 = fluffy pieces with ragged edges/mushy stool, 7 = watery, no solid pieces).
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 21 as determined by stool consistency as per the Bristol Stool Scale | 21 days
  Bristol Stool Scale is a seven-stool description and image scale within the Daily Bowel Habit Diary to assess stool shape and consistency (1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = like a sausage but with cracks on its surface, 4 = like a sausage or snake, smooth and soft, 5 = soft blobs with clear-cut edges, 6 = fluffy pieces with ragged edges/mushy stool, 7 = watery, no solid pieces).
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 7 as determined by gastrointestinal symptoms as per the Gastrointestinal Symptom Rating Scale | 7 days
  The GSRS is a validated, self-assessed, disease-specific scale that will be administered at all in-clinic visits. Five symptom clusters depicted as Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation will be assessed from the combination of the 15 items in the questionnaire (Abdominal pains, Heartburn, Acid regurgitation, Sucking sensations in the epigastrium, Nausea and vomiting, Borborygmus, Abdominal distension, Eructation, Increased flatus, Decreased passage of stools, Increased passage of stools, Loose stools, Hard Stools, Urgent need for defecation, Feeling of incomplete evacuation). All the domains will be scored on a 3-point scale where 1 represented no symptoms and 3 represented severe symptoms
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 14 as determined by gastrointestinal symptoms as per the Gastrointestinal Symptom Rating Scale | 14 days
  The GSRS is a validated, self-assessed, disease-specific scale that will be administered at all in-clinic visits. Five symptom clusters depicted as Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation will be assessed from the combination of the 15 items in the questionnaire (Abdominal pains, Heartburn, Acid regurgitation, Sucking sensations in the epigastrium, Nausea and vomiting, Borborygmus, Abdominal distension, Eructation, Increased flatus, Decreased passage of stools, Increased passage of stools, Loose stools, Hard Stools, Urgent need for defecation, Feeling of incomplete evacuation). All the domains will be scored on a 3-point scale where 1 represented no symptoms and 3 represented severe symptoms
The difference between probiotic and placebo groups in gastrointestinal health from baseline to day 21 as determined by gastrointestinal symptoms as per the Gastrointestinal Symptom Rating Scale | 21 days
  The GSRS is a validated, self-assessed, disease-specific scale that will be administered at all in-clinic visits. Five symptom clusters depicted as Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation will be assessed from the combination of the 15 items in the questionnaire (Abdominal pains, Heartburn, Acid regurgitation, Sucking sensations in the epigastrium, Nausea and vomiting, Borborygmus, Abdominal distension, Eructation, Increased flatus, Decreased passage of stools, Increased passage of stools, Loose stools, Hard Stools, Urgent need for defecation, Feeling of incomplete evacuation). All the domains will be scored on a 3-point scale where 1 represented no symptoms and 3 represented severe symptoms
The change in fecal zonulin levels from baseline to day 7 | 7 days
  Zonulin levels will be analysed from stool samples. A decrease in zonulin levels are associated with better intestinal health.
The change in fecal zonulin levels from baseline to day 14 | 14 days
  Zonulin levels will be analysed from stool samples. A decrease in zonulin levels are associated with better intestinal health.
The change in fecal zonulin levels from baseline to day 21 | 21 days
  Zonulin levels will be analysed from stool samples. A decrease in zonulin levels are associated with better intestinal health.
The change in fecal zonulin levels from baseline to day 28 | 28 days
  Zonulin levels will be analysed from stool samples. A decrease in zonulin levels are associated with better intestinal health.
The change in fecal calprotectin levels from baseline to day 28 | 28 days
  Calprotectin levels will be analysed from stool samples. A decrease in calprotectin levels are associated with better intestinal health.
The change in probiotic impact questionaire from baseline to day 14 | 14 days
  This 22-item questionnaire was specifically designed capture the impact of Lactobacillus plantarum 276 (Lp276) on participants health
The change in probiotic impact questionaire from baseline to day 28 | 28 days
  This 22-item questionnaire was specifically designed capture the impact of Lactobacillus plantarum 276 (Lp276) on participants health
The change in fecal microbial composition from baseline to day 7 | 7 days
  Microbial composition will be analysed from stool samples
The change in fecal microbial composition from baseline to day 14 | 14 days
  Microbial composition will be analysed from stool samples
The change in fecal microbial composition from baseline to day 21 | 21 days
  Microbial composition will be analysed from stool samples
The change in fecal microbial composition from baseline to day 28 | 28 days
  Microbial composition will be analysed from stool samples

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events following 28-day supplementation | 28 days
Change in systolic blood pressure following a 28-day supplementation | 28 days
Change in diastolic blood pressure following a 28-day supplementation | 28 days
Change in heart rate following a 28-day supplementation | 28 days
Change in alanine aminotransferase (ALT) levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in aspartate aminotransferase (AST) levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in total bilirubin levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in creatinine levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in sodium electrolyte levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in potassium electrolyte levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in chloride electrolyte levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in estimated glomerular filtration rate (eGFR) levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in white blood cell count following a 28-day supplementation | 28 days
  Analysed from blood
Change in neutrophil count following a 28-day supplementation | 28 days
  Analysed from blood
Change in lymphocyte count following a 28-day supplementation | 28 days
  Analysed from blood
Change in monocyte count following a 28-day supplementation | 28 days
  Analysed from blood
Change in eosinophil count following a 28-day supplementation | 28 days
  Analysed from blood
Change in basophil count following a 28-day supplementation | 28 days
  Analysed from blood
Change in red blood cell (RBC) count following a 28-day supplementation | 28 days
  Analysed from blood
Change in hemoglobin levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in hematocrit levels following a 28-day supplementation | 28 days
  Analysed from blood
Change in platelet count following a 28-day supplementation | 28 days
  Analysed from blood
Change in mean platelet volume (MPV) following a 28-day supplementation | 28 days
  Analysed from blood
Change in mean corpuscular volume (MCV) following a 28-day supplementation | 28 days
  Analysed from blood
Change in mean corpuscular hemoglobin (MCH) following a 28-day supplementation | 28 days
  Analysed from blood
Change in mean corpuscular hemoglobin concentration (MCHC) following a 28-day supplementation | 28 days
  Analysed from blood
Change in red cell distribution width (RDW) following a 28-day supplementation | 28 days
  Analysed from blood

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No